CLINICAL TRIAL: NCT04835935
Title: The Association Between Milk Feedings in the Preterm Population, the Microbiome and Risk of Atopic Disease
Brief Title: Microbiome, Atopic Disease, Prematurity
Acronym: MAP
Status: Active, not recruiting | Type: Observational
Sponsor: Sydney Leibel (Other)
Responsible Party: Sponsor-Investigator, Sydney Leibel, Assoc Physician, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 181711
Record Dates: First submitted 2021-03-02; First posted 2021-04-08 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Atopy; Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, breast milk, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- subject who developed atopic disease
  Interventions: Other: microbiome pattern
- subject who did not develop atopic disease
  Interventions: Other: microbiome pattern

INTERVENTIONS:
Other: microbiome pattern — microbiome pattern in neonatal period

SUMMARY:
There is increasing recognition that the microbiome may be important in the development of allergic disease. Asthma is the most prevalent pediatric chronic disease and affects more than 300 million people worldwide. For unclear reasons, those infants born at 34 weeks and earlier are three times as likely to develop asthma. Factors such as formula feeding, C-section delivery and antibiotic exposure may play a role. Recent evidence has identified a "critical window" in early life where gut and breast milk microbial changes are most influential. The investigators propose a novel study to follow a cohort of premature babies in the NICU and after discharge home. The investigators aim to examine whether various exposures of babies in the NICU impact their milk and gut microbiome and lead to asthma and allergies.

Our specific aims are:

1. To assess if there is a specific pattern of gut and/or breast milk microbiome over time that is affected by the type of nutrition a baby receives (donor vs maternal vs formula) or other exposures such as antibiotics.
2. Assess whether there are patterns in the microbiome associated with the development of allergic sensitization patterns.
3. Determine if early patterns of the microbiome and allergic sensitization predict allergic conditions (food allergies, allergic rhinitis, eczema, asthma) by 2 years of age.

The investigators will recruit approximately 50 subjects born at 34 weeks of gestation or earlier from two local level III NICU. These subjects will be followed over their NICU course with weekly stool, milk feed, and oral saliva collection as well as documentation of relevant events including prenatal history, delivery history, nutrition and breast feeding history and antibiotic courses. Further samples will be collected after discharge at research visits that will take place Rady Children's Hospital until 4-6 years of age. At these visits, standardized allergy questionnaires and a blood allergy panel will be obtained. Together this data will provide a unique opportunity to identify potential shifts in the microbiome associated with nutrition, asthma and allergy in preterm infants. Ultimately, the investigators may be able to discover ways to prevent the development of asthma and allergies during this early window of opportunity.

ELIGIBILITY:
Inclusion Criteria:

* premature infant equal or less than 34 weeks of age

Exclusion Criteria:

* hypoxic ischemic encephalopathy, congenital anomaly that affects gastrointestinal system, unable to follow up

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants born at equal or less than 34 weeks gestational age.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Atopic Disease | 2-3 years of age
  Clinical diagnosis of any atopic disease among the participants during study follow up visit. These include any food allergies, allergic rhinitis, eczema, and asthma.

SECONDARY OUTCOMES:
Allergic sensitization patterns | 1-2 years
  Allergic sensitization patterns among the participants will be measured by ImmunoCAP Multitest, which is a blood test that provides qualitative responses (positive or negative) for food and environmental allergens.

OTHER OUTCOMES:
Gut, oral and milk feed microbiome | birth to 1 year of age
  Longitudinal stool, oral swab and milk feed samples will be analyzed for paired microbiome and metabolome patterns. The bacterial and metabolomic profiles will be correlated with the allergic sensitization patterns and diagnosis of pediatric atopic disease in participants.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Scripps Memorial Hospital - Rady NICU, San Diego, California
  - University of California, San Diego - Jacobs NICU, San Diego, California

IPD SHARING:
Plan to Share IPD: No
de-identified microbiome and metabolome data will be available.

REFERENCES:
- [Background] Raciborski F, Tomaszewska A, Komorowski J, Samel-Kowalik P, Bialoszewski AZ, Walkiewicz A, Lusawa A, Szymanski J, Opoczynska D, Druzba M, Borowicz J, Lipiec A, Kapalczynski WJ, Samolinski B. The relationship between antibiotic therapy in early childhood and the symptoms of allergy in children aged 6-8 years - the questionnaire study results. Int J Occup Med Environ Health. 2012 Sep;25(4):470-80. doi: 10.2478/S13382-012-0056-0. Epub 2012 Dec 3. PMID 23212289
- [Background] Silvers KM, Frampton CM, Wickens K, Pattemore PK, Ingham T, Fishwick D, Crane J, Town GI, Epton MJ; New Zealand Asthma and Allergy Cohort Study Group. Breastfeeding protects against current asthma up to 6 years of age. J Pediatr. 2012 Jun;160(6):991-6.e1. doi: 10.1016/j.jpeds.2011.11.055. Epub 2012 Jan 30. PMID 22289356
- [Background] Roduit C, Scholtens S, de Jongste JC, Wijga AH, Gerritsen J, Postma DS, Brunekreef B, Hoekstra MO, Aalberse R, Smit HA. Asthma at 8 years of age in children born by caesarean section. Thorax. 2009 Feb;64(2):107-13. doi: 10.1136/thx.2008.100875. Epub 2008 Dec 3. PMID 19052046
- [Background] Been JV, Lugtenberg MJ, Smets E, van Schayck CP, Kramer BW, Mommers M, Sheikh A. Preterm birth and childhood wheezing disorders: a systematic review and meta-analysis. PLoS Med. 2014 Jan 28;11(1):e1001596. doi: 10.1371/journal.pmed.1001596. eCollection 2014 Jan. PMID 24492409
- [Background] Lynch SV, Wood RA, Boushey H, Bacharier LB, Bloomberg GR, Kattan M, O'Connor GT, Sandel MT, Calatroni A, Matsui E, Johnson CC, Lynn H, Visness CM, Jaffee KF, Gergen PJ, Gold DR, Wright RJ, Fujimura K, Rauch M, Busse WW, Gern JE. Effects of early-life exposure to allergens and bacteria on recurrent wheeze and atopy in urban children. J Allergy Clin Immunol. 2014 Sep;134(3):593-601.e12. doi: 10.1016/j.jaci.2014.04.018. Epub 2014 Jun 4. PMID 24908147
- [Background] Arrieta MC, Stiemsma LT, Dimitriu PA, Thorson L, Russell S, Yurist-Doutsch S, Kuzeljevic B, Gold MJ, Britton HM, Lefebvre DL, Subbarao P, Mandhane P, Becker A, McNagny KM, Sears MR, Kollmann T; CHILD Study Investigators; Mohn WW, Turvey SE, Finlay BB. Early infancy microbial and metabolic alterations affect risk of childhood asthma. Sci Transl Med. 2015 Sep 30;7(307):307ra152. doi: 10.1126/scitranslmed.aab2271. PMID 26424567
- [Background] Jeurink PV, van Esch BC, Rijnierse A, Garssen J, Knippels LM. Mechanisms underlying immune effects of dietary oligosaccharides. Am J Clin Nutr. 2013 Aug;98(2):572S-7S. doi: 10.3945/ajcn.112.038596. Epub 2013 Jul 3. PMID 23824724
- [Background] Neu J. Preterm infant nutrition, gut bacteria, and necrotizing enterocolitis. Curr Opin Clin Nutr Metab Care. 2015 May;18(3):285-8. doi: 10.1097/MCO.0000000000000169. PMID 25807349
- [Derived] Luskin K, Mortazavi D, Bai-Tong S, Bertrand K, Chambers C, Schulkers-Escalante K, Ahmad A, Luedtke S, O'Donoghue AJ, Ghassemian M, Geng B, Leibel SL, Leibel SA. Allergen Content and Protease Activity in Milk Feeds from Mothers of Preterm Infants. Breastfeed Med. 2022 Nov;17(11):947-957. doi: 10.1089/bfm.2022.0115. Epub 2022 Oct 12. PMID 36251466